CLINICAL TRIAL: NCT01678222
Title: The Role of Functionally Relevant Cyclooxygenase-2 (COX-2) Gene Single Nucleotide Polymorphisms - 765G>C and 8473T>C in Lymphocyte Differentiation
Brief Title: The COX-2 Gene and the Immune System
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120190; 12-E-0190
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-09-18

CONDITIONS: Allergic Inflammation; Asthma
Keywords: Lymphocyte; Prostaglandin Endoperoxidase Synthase 2; COX-2; Natural History
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SNP: individuals who are homozygous for either the major or minor variant of both SNPs

SUMMARY:
Background:

- The immune system contains several different types of cells in the blood and other parts of the body. The body can fight infections well with the right balance of these cell types. The wrong balance of cell types may cause diseases, such as allergies or asthma. The COX-2 gene may help decide the balance of cell types that the body makes as part of the immune system. It may also play a role in certain immune system diseases. Researchers want to see how COX-2 affects the cells in the immune system.

Objectives:

- To study how the COX-2 gene works in the body s immune system.

Eligibility:

- Individuals 18 years of age and above who are part of the Environmental Polymorphisms Registry.

Design:

* Participants will have one study visit at the National Institutes of Health. They will collect a urine sample at home on the morning of the study visit.
* Participants will have a physical exam and medical history. They will provide a blood sample. They will also give researchers the urine sample they collected that morning.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
This is a cross-sectional, controlled study designed to investigate the association of single nucleotide polymorphisms (SNPs) in the cyclooxygenase-2 (COX2) gene, also called prostaglandin endoperoxidase synthase 2 (PTGS2), on T-cell differentiation and function. Specifically, the impact of the promoter-region SNP 765G>C (rs20417) and the 3 untranslated region (UTR) SNP 8473T>C (rs5275) on T helper cell (Th) 2, Th9, and Th17 differentiation and function will be examined. Non-Hispanic, White or Black/African American, non-pregnant adults, aged 18-65 years, who are wild type (WT), with respect to both the 765G>C and 8473T>C SNPs, WT with respect to 765G>C and homozygous for 8473T>C, and homozygous for both 765G>C and 8473T>C will be recruited into a total of three genotype groups. Potential participants will be identified from the Environmental Polymorphisms Registry, contacted by recruitment letter and pre-screened for eligibility. Pre-screened individuals will provide verbal consent to withhold certadata analysis, a urine collection cup, and pre-visit instructions. Participants will attend a single study visit that will take place at the National Institute of Environmental Health Sciences (NIEHS) Clinical Research Unit (CRU). During this visit, written informed consent will be obtained, and there will be a final screening and eligibility determination, medical history review, vital signs, physical examination and blood and urine samples will be collected. From peripheral blood, lymphocyte subsets, prostaglandin levels, and cytokine levels will be determined; stable prostaglandin metabolites, creatinine, total protein and albumin will be measured in urine. Lymphocytes will be isolated from peripheral blood for ex vivo analyses. Demographic characteristics (i.e., age) will be compared between the groups, and when possible, recruitment will be targeted to achieve an approximate match of race and gender across the groups. The primary objective of the study is to determine whether the 765G>C or 8473T>C SNPs exhibit altered Th2, Th9 and Th17 cell differentiation by examining lymphocyte subsets in vivo. The study will also examine the impact of these two SNPs on circulating Th2/Th9/Th17 cytokine levels and prostaglandins in vivo, on differentiation of naive CD4+T-cells to Th cell subsets in vitro, and on lymphocyte production of cytokines and prostaglandins in vitro.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant of the Environmental Polymorphisms Registry and current contact information available
* Genotype information available for relevant 765G>C and 8473T>C COX2 polymorphisms, which indicates:

  * Individuals who are WT with respect to both 765G>C and 8473T>C (N=31)
  * Individuals who are WT with respect to 765G>C and homozygous for 8473T>C (N=31)
  * Individuals who are homozygous for both 765G>C and 8473T>C (N=31)
* Age 18- 65 years
* Race self-identified as White or Black and Non-Hispanic ethnicity
* Willing and able to provide informed consent
* Able to comply with all protocol procedures

EXCLUSION CRITERIA:

* History of infection within the preceding 1 week or an oral temperature >38 degrees C
* Current daily or chronic use of corticosteroids (systemic, inhaled and topical).
* Any current conditions known to impact peripheral white blood cell count (e.g., leukemia, lymphopenia, AIDS, other immunodeficiency disorders)
* Current daily or chronic use of systemic immunosuppressants.
* Current pregnancy or lactation
* Unwilling or unable to:

  * Fast (including alcohol and caffeine-containing products) and discontinue tobacco use for 12 hours prior to the study visit
  * Withhold all prescribed and over-the-counter medications and supplements the morning of the study visit, until after the visit is completed
  * Refrain from taking the following medications and supplements for 7 days prior to the study visit:

    * NSAIDs
    * Corticosteroids (nasal, inhaled, topical or systemic)
    * Fish oil and niacin supplements
* For blood draws that exceed 200ml, a hematocrit of <34% for women or <36% for men, or >56% for either gender.
* For blood draws exceeding 200ml, blood or plasma donation in the last 8 weeks

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals who are homozygous for either the major or minor variant of both SNPs@@@
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2013-05-02 (Actual)

PRIMARY OUTCOMES:
To determine whether 765>C is associated with altered Th2, Th9, and Th17 differentiation in vivo | Ongoing
  To determine whether 765>C is associated with altered Th2, Th9, and Th17 differentiation in vivo
To determine whether 8473T>C is associated with altered Th2, Th9, and Th17 differentiation in vivo | Ongoing
  To determine whether 8473T>C is associated with altered Th2, Th9, and Th17 differentiation in vivo

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Li H, Bradbury JA, Dackor RT, Edin ML, Graves JP, DeGraff LM, Wang PM, Bortner CD, Maruoka S, Lih FB, Cook DN, Tomer KB, Jetten AM, Zeldin DC. Cyclooxygenase-2 regulates Th17 cell differentiation during allergic lung inflammation. Am J Respir Crit Care Med. 2011 Jul 1;184(1):37-49. doi: 10.1164/rccm.201010-1637OC. Epub 2011 Apr 7. PMID 21474648
- [Background] McAdam BF, Catella-Lawson F, Mardini IA, Kapoor S, Lawson JA, FitzGerald GA. Systemic biosynthesis of prostacyclin by cyclooxygenase (COX)-2: the human pharmacology of a selective inhibitor of COX-2. Proc Natl Acad Sci U S A. 1999 Jan 5;96(1):272-7. doi: 10.1073/pnas.96.1.272. PMID 9874808
- [Background] Mai J, Wang H, Yang XF. Th 17 cells interplay with Foxp3+ Tregs in regulation of inflammation and autoimmunity. Front Biosci (Landmark Ed). 2010 Jun 1;15(3):986-1006. doi: 10.2741/3657. PMID 20515737
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-E-0190.html